CLINICAL TRIAL: NCT03881735
Title: A Phase II Study of Intensive Salvage Therapy Followed by Enasidenib for Patients With AML Harboring Mutations in IDH2 Who Have Failed or Been Refractory to One Prior Line of Therapy
Brief Title: Enasidenib in Treating Patients With Relapsed or Refractory Acute Myeloid Leukemia With an IDH2 Gene Mutation
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: no accrual
Sponsor: Roswell Park Cancer Institute (Other)
Collaborators: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: I 67118; NCI-2019-00332 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); I 67118 (Other: Roswell Park Cancer Institute)
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Blasts Under 5 Percent of Peripheral Blood White Cells; Bone Marrow Blasts Decreased by 50 Percent or More Compared to Pretreatment Level; IDH2 Gene Mutation; Recurrent Acute Myeloid Leukemia; Refractory Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — enasidenib; Stem Cell Transplantation; Hematopoietic Stem Cell Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort A (enasidenib, hematopoietic cell transplantation) (Experimental): Patients receive enasidenib PO QD. Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo a HCT 7-14 days after treatment. Within 30-100 days following the transplant, patients receive enasidenib QD. Treatment repeats every 28 days for 24 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enasidenib; Procedure: Hematopoietic Cell Transplantation
- Cohort B (enasidenib) (Active Comparator): Patients receive enasidenib PO QD. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Enasidenib

INTERVENTIONS:
Drug: Enasidenib — Given PO
  Other Names: AG-221; CC-90007
Procedure: Hematopoietic Cell Transplantation — Undergo HCT
  Other Names: HCT; Hematopoietic Stem Cell Transplantation; HSCT; stem cell transplantation
  Arms: Cohort A (enasidenib, hematopoietic cell transplantation)

SUMMARY:
This phase II trial studies how well enasidenib works in treating in patients with acute myeloid leukemia with an IDH2 gene mutation that has come back or has not responded to treatment. Enasidenib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. In this study we are investing if enasidenib can be used as maintenance therapy post salvage induction chemotherapy.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the effect of IDH2 inhibition following conventional high dose salvage chemotherapy with detectable IDH2 mutations on event free survival (EFS) in patients with relapsed/refractory acute myeloid leukemia (AML).

SECONDARY OBJECTIVES:

I. Evaluate the effect of IDH2 inhibitor maintenance therapy following intensive salvage therapy: i.e., rate of hematocrit (HCT), duration of maintenance therapy and overall survival in patients with IDH2 mutant relapsed/refractory AML.

EXPLORATORY OBJECTIVES:

I. Evaluate the changes in IDH2 mutational variant allelic frequency and deoxyribonucleic acid (DNA) methylation signature while on enasidenib therapy.

OUTLINE: Patients are assigned to 1 of 2 cohorts.

COHORT I: Patients receive enasidenib orally (PO) once daily (QD). Treatment repeats every 28 days for up to 6 cycles in the absence of disease progression or unacceptable toxicity. Patients then undergo a hematopoietic cell transplantation (HCT) 7-14 days after treatment. Within 30-100 days following the transplant, patients receive enasidenib QD. Treatment repeats every 28 days for 24 cycles in the absence of disease progression or unacceptable toxicity.

COHORT II: Patients receive enasidenib PO QD. Treatment repeats every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 6 months and then yearly for 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of AML harboring a mutation in IDH2 relapsed or refractory to first line cytarabine/anthracycline induction chemotherapy, failed to respond to or relapsed following at least 2 cycles of hypomethylating agent (azacitidine, decitabine, sgi-110) or at least 1 cycle of hypomenthylating agent with venetoclax or other targeted therapies

  * Patients will be identified and deemed eligible based upon the identification of an IDH2 mutation identified at either at the time of disease relapse prior to re-induction chemotherapy or following 1-2 cycles of chemotherapy induction. Each institution will test using their standard local FDA-approved or cleared assay per the institutional standard of care workup for relapsed disease.
  * First relapse defined as untreated hematologic relapse (according to International Working Group criteria) after one line of intensive regimen for AML including at least one cytarabine containing induction block with a total dose no less than 700 mg/m^2 per cycle and 3 days of an anthracycline that induced a complete remission (CR)/complete remission with incomplete hematologic recovery (CRi)/complete remission with incomplete platelet recovery (CRp). Subjects are allowed to receive induction, consolidation, transplant and/or maintenance therapy prior to achieving their first CR/CRi/CRp
  * Refractory to induction therapy is defined as never achieving CR, CRi or CRp (according to International Working Group criteria) after one line of intensive regimen for AML (reinduction, consolidation and/or transplant allowed) including at least one cytarabine containing induction block with a total dose no less than 700 mg/m^2 per cycle and 3 days of an anthracycline
* Subjects considered eligible for intensive chemotherapy
* Subjects had received a first salvage within the last 60 days (day 15 to 60 following most recent cytarabine-based standard salvage number [#] 1 therapy) who achieved either > 50% reduction in blast percentage from the pre-treatment bone marrow OR < 20% cellularity with any blast percentage AND < 5% peripheral blood blasts
* Have an Eastern Cooperative Oncology Group (ECOG) performance status of =< 2
* Adequate liver function within 72 hours of enrollment, defined as:

  o Blood total bilirubin ≤ 1.5 x ULN, unless considered due to Gilbert's syndrome (eg, a gene mutation in UGT1A1) or leukemic organ involvement, following review by the Investigator
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3.0 x upper limit of normal (ULN) (within 72 hours of enrollment)
* Adequate renal function within 72 hours of enrollment, defined as blood creatinine =< 2.5 x ULN
* Females of childbearing potential (FCBP) may participate, providing they meet the following conditions:

  * Agree to practice true abstinence from sexual intercourse or to use highly effective contraceptive methods (eg, combined [containing estrogen and progestogen] or progestogen-only associated with inhibition of ovulation, oral, injectable, intravaginal, patch, or implantable hormonal contraceptive; bilateral tubal occlusion; intra-uterine device; intrauterine hormone-releasing system; or male partner sterilization [note that vasectomized partner is a highly effective birth control method provided that partner is the sole sexual partner of the FCBP trial participant and that the vasectomized partner has received medical assessment of the surgical success]) at screening and throughout the study, and for 4 months following the last study treatment (6 months following the last dose of cytarabine); and
  * Have a negative serumblood β-subunit of human chorionic gonadotropin (β-hCG) pregnancy test (sensitivity of at least 25 mIU/mL) at screening; and
  * Have a negative serum or urine (investigator's discretion under local regulations) β hCG pregnancy test (sensitivity of at least 25 mIU/mL) within 72 hours prior to the start of study treatment in the Treatment Phase (note that the screening serumblood pregnancy test can be used as the test prior to the start of study treatment in the Treatment Phase if it is performed within the 72 hour timeframe).
* Men must use a latex condom during any sexual contact with women of childbearing potential
* Willing to adhere to protocol specific requirements
* Clinically significant toxic effects of prior therapy (except hydroxyurea) resolved to grade =< 1 before the start of study
* Participant or legal representative must understand the investigational nature of this study and sign an Independent Ethics Committee/Institutional Review Board approved written informed consent form prior to receiving any study related procedure

Exclusion Criteria:

* Acute promyelocytic leukemia (APL)
* Subject has or is suspected of having central nervous system (CNS) leukemia. Evaluation of cerebrospinal fluid is only required if CNS involvement by leukemia is suspected during screening
* Clinically active or unstable graft-versus-host disease (GVHD) requiring treatment that precludes administration of chemotherapy as defined in this protocol
* Prior anti-leukemia therapy within 5 x the half-life for other investigational agents

  * Prior use of hydroxyurea or isolated doses of cytarabine for palliation (i.e., control of white blood count [WBC]) are allowed but should be discontinued at least 24 hours prior to enrollment. Other agents used strictly with palliative intent might be allowed during this period after discussing with principal investigator
* Pre-existing liver disease (e.g. cirrhosis, chronic hepatitis B or C, nonalcoholic steatohepatitis, sclerosing cholangitis)
* Subject is known seropositive or active infection with human immunodeficiency virus (HIV), or active infection with hepatitis B virus (HBV) or hepatitis C virus (HCV)
* Subject has active uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics, antiviral therapy, and/or other treatment)
* Pregnant or nursing female participants
* Subjects of childbearing potential not willing to use adequate contraception
* Subject has significant active cardiac disease within 6 months prior to the start of study treatment, including New York Heart Association (NYHA) class III or IV congestive heart failure; acute coronary syndrome (ACS); and/or stroke; or left ventricular ejection fraction (LVEF) < 40% by echocardiogram (ECHO) or multi-gated acquisition (MUGA) scan obtained within 28 days prior to the start of study treatment
* Subject with concurrent severe and/or uncontrolled medical or psychiatric conditions that in the opinion of the investigator may impair the participation in the study or the evaluation of safety and/or efficacy
* Subject has immediately life-threatening, severe complications of leukemia such as uncontrolled bleeding, pneumonia with hypoxia or shock, and/or disseminated intravascular coagulation
* Subject is known to have dysphagia, short-gut syndrome, gastroparesis, or other conditions that limit the ingestion or gastrointestinal absorption of drugs administered orally
* Subjects has uncontrolled hypertension (systolic blood pressure [BP] > 180 mmHg or diastolic BP > 90 mmHg)
* Subject has known (or suspected to have) hypersensitivity to any of the components of study treatment
* Subject has corrected QT (QTc) interval (i.e., Fridericia's correction [QTcF]) >= 450 ms or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome) at screening
* Subject is taking the following sensitive CYP substrate medications that have a narrow therapeutic range are excluded from the study unless the subject can be transferred to other medications at least 5 half-lives prior to the start of study treatment: phenytoin (CYP2C9), S-mephenytoin (CYP2C19), thioridazine (CYP2D6), theophylline, and tizanidine (CYP1A2)
* Subject who is taking the breast cancer resistance protein (BCRP) transporter-sensitive substrate (i.e., rosuvastatin) should be excluded from the study unless the subject can be transferred to other medications at least 5 half-lives prior to the start of study treatment
* Subject with prior history of malignancy, other than myelodysplastic syndrome (MDS), myeloproliferative neoplasm (MPN) or AML may be eligible after discussion with the study doctor. Diagnoses of basal or squamous cell carcinoma of the skin, carcinoma in situ of the cervix, carcinoma in situ of the breast, and previously treated prostate cancer (T1a/T1b by TNM staging) are not exclusionary :
* Concurrent participation in another therapeutic clinical trial
* Unwilling or unable to follow protocol requirements
* Any condition which in the investigator's opinion deems the participant an unsuitable candidate to receive study drug Subject has any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-12-02 (Actual); Primary Completion 2021-11-19 (Estimated); Study Completion 2022-11-19 (Estimated)

PRIMARY OUTCOMES:
Event-free survival (EFS) in each cohort | At 12 months
  Defined as the binomial proportion of evaluable patients who are alive and disease free 12 months after enrollment. Two-sided 95% Jeffreys confidence interval estimates will be used to describe the plausible range for the true EFS rate in each patient group. The EFS rates will be estimated separately for each cohort, on an intent-to-treat basis.

SECONDARY OUTCOMES:
Success rate of hematopoietic cell transplantation (HCT) | Up to 5 years
Median duration of maintenance therapy in both cohorts | Up to 5 years
Overall survival in each cohort | At 12 and 24 months

OTHER OUTCOMES:
Evaluation of IDH2 mutant allele burden | Up to 5 years
  Will use droplet digital polymerase chain reaction (PCR) from baseline study entry and at follow up every 3 months to follow changes in variant allele frequency (VAF).
Change in deoxyribonucleic acid (DNA) methylation signature | Up to 5 years
  Will be evaluated by evaluated by bi-sulfite pyrosequencing.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Griffiths, MD, Principal Investigator — Roswell Park Cancer Institute
Locations (2):
- United States (2):
  - Roswell Park Cancer Institute, Buffalo, New York
  - Cancer Institute at St Francis Hosptial, East Hills, New York